CLINICAL TRIAL: NCT05311150
Title: A Randomized Control Trial to Compare the Diagnostic Yield of Endobronchial Biopsy Performed Under Direct Narrow Band Imaging or White Light Bronchoscopy Guidance in Suspected Sarcoidosis
Brief Title: An RCT of NBI vs. White Light Guided Endobronchial Biopsy in Suspected Sarcoidosis
Acronym: NABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Associate Professor of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INT/IEC/2021/SPL-1817
Record Dates: First submitted 2022-03-26; First posted 2022-04-05 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Masking Description: The pathologist analyzing the biopsy specimen will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrow band imaging bronchoscopy (Active Comparator): The narrow band imaging mode uses two narrow bands of light with wavelengths of 390-445 nm and 530-550 nm.
  Interventions: Device: Narrow band imaging bronchoscopy guided endobronchial biopsy
- White light bronchoscopy (Active Comparator): The white light bronchoscopy mode uses the entire range of white light wavelengths, 400-700 nm.
  Interventions: Device: White light bronchscopy guided endobronchial biopsy

INTERVENTIONS:
Device: Narrow band imaging bronchoscopy guided endobronchial biopsy — Examination of the airways will be performed with the narrow band imaging mode using a flexible video-bronchoscope (BF-1T 180, Olympus Medical, Japan). Endobronchial biopsies will be performed from the abnormal areas as deemed by the operator.
  Arms: Narrow band imaging bronchoscopy
Device: White light bronchscopy guided endobronchial biopsy — Examination of the airways will be performed with the white light bronchoscopy mode using a flexible video-bronchoscope (BF-1T 180, Olympus Medical, Japan). Endobronchial biopsies will be performed from the abnormal areas as deemed by the operator.
  Arms: White light bronchoscopy

SUMMARY:
In the diagnosis of patients with sarcoidosis, there is paucity of literature on the diagnostic yield of the endobronchial biopsies obtained with narrow band imaging (NBI) bronchoscopy. The present study aims to compare the diagnostic yield of endobronchial biopsyperformed under direct narrow band imaging or white light bronchoscopy guidance in suspected sarcoidosis.We hypothesize that the use of NBI will improve the yield of endobronchial biopsy in patients with sarcoidosis.

DETAILED DESCRIPTION:
The present study will be a randomized controlled trial. It will be performed in the Bronchoscopy suite of the Department of Pulmonary Medicine, PGIMER. Subjects meeting the selection criteria will be randomized 1:1 to undergo EBB under real-time visualization with NBI or white light bronchoscopy. The randomization sequence will be computer generated and the study group allocations will be placed in opaque sealed envelopes. They will be opened just before the performance of the bronchoscopic procedures.

Primary outcome:the diagnostic yield of EBB (demonstration of granulomatous inflammation in EBB specimen, in subjects with a final diagnosis of sarcoidosis)

Secondary outcomes:

1. Complications related to the procedure (bleeding)
2. Duration of procedure (from the time of entry into the trachea till the completion of the endobronchial biopsy)

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years.
2. Clinical presentation and radiological findings (enlarged hilar and or mediastinal lymph nodes >10 mm [short axis], and/or perilymphatic nodules or peribronchovascular thickening on computed tomography [CT] chest) suggesting sarcoidosis.
3. Willing to give informed consent.

Exclusion Criteria:

1. Hemodynamic instability (systolic BP <100 mm Hg).
2. Pregnancy.
3. Treatment with systemic glucocorticoids for more than three weeks in the preceding three months.
4. Diagnosis of sarcoidosis possible with another minimally invasive technique such as skin biopsy or peripheral lymph node biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Yield of granulomatous inflammation in endobronchial biopsy in subjects with a final diagnosis of sarcoidosis | 7 days
  Diagnostic yield of endobronchial biopsy (demonstration of granulomatous inflammation in EBB specimen, in subjects with a final diagnosis of sarcoidosis)

SECONDARY OUTCOMES:
Complications: Bleeding | 1 day
  The incidence of bleeding after the endobronchial biopsy
Procedure duration | 1 day
  Duration of procedure (from the time of entry into the trachea till the completion of the endobronchial biopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh N Aggarwal, MD, DM, Study Chair — PGIMER, Chandigarh, India
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rathi K, Dogra P, Agarwal R, Singh Sehgal I, Muthu V, Thurai Prasad K, Aggarwal AN, Bal A, Gupta N, Dhooria S. A randomized trial of narrow band imaging for performing airway mucosal biopsy in pulmonary sarcoidosis (NABS). Sarcoidosis Vasc Diffuse Lung Dis. 2025 Sep 30;42(3):16418. doi: 10.36141/svdld.v42i3.16418. PMID 41026031